CLINICAL TRIAL: NCT06800469
Title: Gut Microbiota Analysis in Patients Undergoing Duodencephalopancreasectomy for Pancreatic Cancer (MIcRobiome Analysis in Patients UnderGoing PancrEatico-duodenectomy for Pancreatic Cancer MIRAGE Study)
Brief Title: Gut Microbiota Analysis in Patients Undergoing Duodencephalopancreasectomy for Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIRAGE study
Record Dates: First submitted 2025-01-09; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer, Adult
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic cancer, adult; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with adenocarcinoma of the pancreas (Other): Patients with adenocarcinoma of the pancreas needing surgical treatment by duodenocephalopancreasect
  Interventions: Diagnostic Test: Microbiota analysis

INTERVENTIONS:
Diagnostic Test: Microbiota analysis — Upon acquisition of informed consent, fecal, digiunal mucosa, biliary and pancreatic fluid samples will be collected for microbiota analysis

SUMMARY:
Pancreatic head cancer represents one of the most frequent malignancies with an incidence of about 13500 new cases each year. The primary objective of the study is to test whether there are bacterial species associated with increased risk of complications in patients with peri-ampullary neoplasia undergoing DCP.

DETAILED DESCRIPTION:
Pancreatic head cancer represents one of the most frequent malignancies with an incidence of about 13500 new cases each year. The only curative strategy for such neoplasm is still surgical resection by duodenocephalopancreasectomy (DCP) surgery. However, this procedure has a postoperative morbidity of about 70% with a severe complication rate of 20%. The most frequent complications are pancreatic fistula, biliary fistula, and infectious complications in general. These complications often account for a high postoperative mortality rate that even in high-volume centers reaches 5%. Although some predictive risk factors are known (comorbidities and the patient's age, the consistency of the pancreatic stump to be anastomized and/or type of pathology treated), there is still no study that has evaluated the influence of the gut microbiota in the determinism of complications. This hypothesis appears suggestive and supported by indirect evidence from the literature. Some preliminary studies performed in the field of colo-rectal surgery have shown that the presence of certain bacterial families such as Lachnospiraceae or Bacteroidaceae are correlated with a significant increase in anastomotic dehiscence. Low microbial diversity also appears to be correlated with increased risk of anastomotic dehiscence. In contrast, the presence of other species such as Prevotella copri or Streptococcus genus seem to correlate with a reduced risk of dehiscence.

The primary objective of the study is: to test whether there are bacterial species associated with increased risk of complications in patients with peri-ampullary neoplasia undergoing DCP.

Other objectives to be verified are:

1. the association between bacterial species and the occurrence of pancreatic fistula in terms of frequency and severity
2. the association between bacterial species and the occurrence of biliary fistula in terms of frequency and severity
3. the association between bacterial species and the occurrence of infectious complications of any kind.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of resectable pancreatic adenocarcinoma with indication for "upfront" surgical treatment
* ASA (American Society of Anesthesiology) score < 4
* Obtaining informed consent

Exclusion Criteria:

- Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Structure of the gut microbiome | 7 days before surgery, 15 and 30 days after surgery thereafter
  The structure of the gut microbiome will be characterized on the samples by "next-generation sequencing" of the hypervariable region V3 to V4 of the 16S rRNA gene (bacterial component) and by "shotgun genomics"; ecosystem functionality will be assessed by measuring the fecal concentration of short-chain fatty acids (SCFA).

CONTACTS AND LOCATIONS:
Overall Officials: Ricci Claudio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy